CLINICAL TRIAL: NCT01323348
Title: Effect of Diabetes Education During Retinal Ophthalmology Visits on Diabetes Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DRCR.net-Protocol M
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes; Diabetic Retinopathy
Keywords: Diabetes; Diabetes Education; Diabetic Retinopathy; HbA1c
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetes Educational Intervention (Experimental): Study participants in the intervention group will receive a diabetes management educational intervention at baseline and at follow-up visits. For those on an annual follow-up schedule, educational intervention will take place at baseline and 12 months. For those whose standard care involves more frequent, than annual, visits the educational intervention will take place no more than once every 12 weeks.
  Interventions: Behavioral: Diabetes Education
- Standard Care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Diabetes Education — The intervention will consist of the following at enrollment and at each follow-up visit (but no more frequently than once every 12 weeks):
  * Measurement of HbA1c in office with immediate feedback
  * Measurement of blood pressure with immediate feedback
  * Assessment of retinopathy risk with immediate feedback
  * Personalized risk assessment reports based on current HbA1c
  * Brief assessment of patient understanding of key issues with immediate feedback
  * Supplemental diabetes management educational materials (provided at baseline only)
  * Feedback to primary care provider
  * Email reminder to study participants with email access of individualized risk assessment findings
  Arms: Diabetes Educational Intervention

SUMMARY:
The purpose of this study is to assess whether glycemic control (assessed with HbA1c measurement) in individuals with type 1 or type 2 diabetes can be improved with a point-of-care measurement of HbA1c in the ophthalmologist's office combined with a personalized risk assessment for diabetic retinopathy and other complications of diabetes.

DETAILED DESCRIPTION:
Although each patient with diabetes should be receiving diabetic education as part of their on-going routine medical care, it is likely that such education is delivered with different details and intensity. Motivating a patient with diabetes to become involved in his or her care is of primary importance in achieving better systemic control.

Ocular complications from diabetes remain the most common cause of blindness among American adults 20-74 years of age. A recent survey reported that loss of vision is the most feared of all diabetic complications. Thus, it is possible that an educational intervention at an ophthalmology office may have additional impact beyond the current standard of diabetes education at a primary care or diabetologist/endocrinologist office alone. This study will determine whether diabetes education in the ophthalmology office (which includes same-visit feedback of HbA1c levels, combined with standardized education regarding same-visit blood pressure, retinopathy status and overall diabetes education) can improve subsequent HbA1c as compared with current standard care in an ophthalmology office.

Materials used in this research setting must be applicable for use in ophthalmology practices. Therefore, the materials and procedures for this study have been developed with the goal of easy translation to this audience.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Diagnosis of type 1 or type 2 diabetes mellitus

   Any one of the following will be considered to be sufficient evidence that diabetes is present:
   * Current regular use of insulin for the treatment of diabetes
   * Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes
   * Documented diabetes by American Diabetes Associate and/or World Health Organization criteria
3. Routine care follow-up is yearly or more frequent
4. English or Spanish speaking
5. Able and willing to provide informed consent
6. Willing to complete 24 months of study follow up

Exclusion Criteria:

1. Known HbA1c (patient report or available records at time of enrollment) <7.5% within prior 6 months
2. Active participation in any type of intervention study
3. Initiation of insulin treatment within 3 months from date of enrollment
4. Prior complete panretinal photocoagulation or prior diabetes-related vitrectomy in both eyes
5. Advanced visual acuity loss in both eyes which prohibits ability to read study materials (tested as needed with reading test using materials in appropriate size script)
6. Significant renal disease including use of erythropoietin (Procrit, Epogen, Eprex) or a history of chronic renal failure requiring dialysis or kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1875 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 12 Months
  Mean change in HbA1c from baseline to 12 months in intervention versus control for study participants being seen for standard care more frequently than every 12 months

SECONDARY OUTCOMES:
Diabetes Care Knowledge | 12 Months/24 Months
  At baseline and at annual visits, study participants in all treatment groups will complete self-assessment questionnaires in order to assess perception of emotional problems frequently reported in type 1 and type 2 diabetes and to measure perceived adherence to diabetes self-care recommendations. At the annual visits, summary statistics will be presented on the responses as appropriate to the distribution and the treatment groups will be compared controlling for baseline responses.
Blood Pressure | 12 Months/24 Months
  For analyses, systolic and diastolic blood pressure will be converted to an overall mean blood pressure according to the following calculation: diastolic blood pressure + 1/3 (systolic blood pressure - diastolic blood pressure). Blood pressure will be analyzed as the change in the weighted mean blood pressure from baseline to 12 months adjusted for the baseline weighted mean blood pressure. Treatment group comparisons will be made using ANCOVA to adjust for the baseline blood pressure, with GEE to adjust for the correlation within subjects of the same cluster.
Body Mass Index | 12 Months/24 Months
  Treatment group comparisons will be made using analysis of covariance (ANCOVA) to adjust for the baseline HbA1c, with generalized estimating equations (GEE) to adjust for the correlation within subjects of the same randomization cluster.

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd P Aiello, M.D., Study Chair — Joslin Diabetes Center
Locations (34):
- United States (34):
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - California Retina Consultants, Santa Barbara, California
  - Retina Vitreous Consultants, Fort Lauderdale, Florida
  - University of Florida College of Med., Department of Ophthalmology, Jacksonville, Florida
  - Central Florida Retina Institute, Lakeland, Florida
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - John-Kenyon American Eye Institute, New Albany, Indiana
  - Retina and Vitreous Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Wilmer Ophthalmological Institute at Johns Hopkins, Baltimore, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford Health System, Dept of Ophthalmology and Eye Care Services, Detroit, Michigan
  - Retina Center, PA, Minneapolis, Minnesota
  - Barnes Retina Institute, St Louis, Missouri
  - The New York Eye and Ear Infirmary/Faculty Eye Practice, New York, New York
  - University of North Carolina, Dept of Ophthalmology, Chapel Hill, North Carolina
  - Charlotte Eye, Ear, Nose and Throat Assoc., PA, Charlotte, North Carolina
  - Wake Forest University Eye Center, Winston-Salem, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania
  - Palmetto Retina Center, Columbia, South Carolina
  - Carolina Retina Center, Columbia, South Carolina
  - Retina Research Center, Austin, Texas
  - Retina and Vitreous of Texas, Houston, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin-Madison, Dept of Ophthalmology/Retina Service, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Aiello LP, Ayala AR, Antoszyk AN, Arnold-Bush B, Baker C, Bressler NM, Elman MJ, Glassman AR, Jampol LM, Melia M, Nielsen J, Wolpert HA; Diabetic Retinopathy Clinical Research Network. Assessing the Effect of Personalized Diabetes Risk Assessments During Ophthalmologic Visits on Glycemic Control: A Randomized Clinical Trial. JAMA Ophthalmol. 2015 Aug;133(8):888-96. doi: 10.1001/jamaophthalmol.2015.1312. PMID 25996273
- See also: Related Info — http://www.drcr.net